CLINICAL TRIAL: NCT04928885
Title: Evaluation of the Wits Workout Wellness Program for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Julie L Bobitt, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-0305; P30AG022849 (NIH)
Record Dates: First submitted 2021-05-19; First posted 2021-06-16 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cognitive Decline; Social Isolation; Health Behaviors; Self Efficacy
Keywords: Cognitive Health; Older Adults; Socialization
MeSH Terms: conditions — Cognitive Dysfunction; Social Isolation; Health Behavior

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized trial with a treatment group and a waitlist control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WW Treatment Group (Experimental): Individuals will receive the 12-week Wits Workout Program. Individuals will take the baseline, 3 mos and 6 mos follow-up surveys. They will also take the Wits Workout satisfaction survey and participate in the 6 mos focus-groups.
  Interventions: Behavioral: Wits Workout Program
- WW Control Group (Other): Individuals will be on a waitlist and will take the baseline, 3 mos and 6 mos. assessments. They will receive the Wits Workout workshop after the 6 month study period is completed.
  Interventions: Other: Control Group that receives intervention after the study

INTERVENTIONS:
Behavioral: Wits Workout Program — 12 week, one hour per week multi-modal, interactive training.
  Arms: WW Treatment Group
Other: Control Group that receives intervention after the study — The control group will not receive the intervention during study period but will take baseline, 3 mos and 6 mos surveys. They will complete the workshop after the study period is over.
  Arms: WW Control Group

SUMMARY:
About 11% of the U.S. older adult population is at risk for or suffers from subjective cognitive decline. While some factors such as genetics and habitual physiological changes that affect brain health cannot be changed, research has shown that lifestyle changes such as participation in regular physical activity, staying socially engaged, and managing stress and diet can help to delay or reduce cognitive decline. Yet few brain health promotion programs exist and those that do fail to focus on global health and wellness as a strategy to improve brain health. Wits Workout is a holistic, 12-session, 60-minute per session, multi-modal workshop series that offers adults ages 50 and older facilitated, interactive dialogue and activities about behaviors that promote brain health. Each week includes a different themed module which has four activities and a training component.

DETAILED DESCRIPTION:
While research has shown that lifestyle changes such as participation in regular physical activity, staying socially engaged, and managing stress can help to delay or reduce cognitive decline, few cognitive brain health programs exist. Those that do are targeted to a specific audience (i.e., Alzheimer's and related dementias) and primarily focus on one health domain (i.e. physical activity, diet) without the additional focus on multi-dimensions of health, which can also include intellectual engagement, social isolation, stress, sleep, and self-efficacy. Thus, there is a need for a more holistic cognitive health program aimed toward the general older adult population and particularly those that are underserved due to geographic location.

Wits Workout, is a multi-modal 12-session (60 min/week) workshop series designed to enhance brain health among people ages 50 and older. Wits Workout addresses multiple factors that affect cognitive health such as physical activity, diet, intellectual engagement, social isolation, stress, sleep, and self-efficacy. The holistic workshop series is designed to be lay-leader led, interactive, and experiential. Preliminary evaluations demonstrate that this educational series serves a need in reducing isolation, increasing physical activity, promoting intellectual engagement, and enhancing overall brain health in older participants, all of which complement current aging brain health research. The researchers propose to conduct a two-arm randomized controlled trial with a treatment (workshop) group (n=120) and wait-list control group (n=120) who will receive the program after the 6-month study period is completed.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older
* English-speaking and/or able to understand English
* Have no diagnosis of Alzheimer's or related dementia
* Score 28 or higher on the TICS cognitive screening
* Able to participate in the 12 week program
* Have not previously participated in a Wits Workout program

Exclusion Criteria:

* Under age 50,
* Unable to speak or understand English,
* Have a diagnosis of Alzheimer's or related dementia,
* Score lower than 28 on TICS
* Plan to miss more than two weeks of the program (i.e. traveling during that time period)
* Have previously participated in a Wits Workout program.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Bobitt, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WW Treatment Group | WW Control Group
Started | 152 | 133
3 Months | 130 | 123
Completed | 123 | 122
Not Completed | 29 | 11

BASELINE CHARACTERISTICS:
Population: Loss to follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | WW Treatment Group | WW Control Group | Total
Number analyzed (Participants) | 152 | 133 | 285
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.05921053 (10.24936345) | 65.03759398 (8.82438599) | 65.58246 (9.607676)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 121 | 257
  Male | 16 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 146 | 126 | 272
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 8 | 22
  White | 134 | 119 | 253
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 152 | 133 | 285

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function
Description: The PROMIS Cognitive Function measure used to measure cognitive functioning. Raw score is converted into the T-score, with 50 being the mean score. 10 T-score is one standard deviation. Therefore, score above 50 means that a person is better than the average population in mental ability, and lower score meaning worse or disability. The score changing over time can indicate decline in cognitive function (lower score) or improved cognitive function (higher score) or no decline or improvement (same score).
Time Frame: Baseline prior to the workshop, at 3 months after baseline and at 6 months after baseline
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | WW Treatment Group | WW Control Group
Number analyzed (Participants) | 130 | 123
T score
  3 Months | 0.28 (4.27) | .65 (4.08)
  6 Months: number analyzed (Participants) | 123 | 122
  6 Months | 1.84 (7.93) | -.73 (6.97)

2. Primary Outcome: Change in Cognitive Status
Description: Telephone Interview for Cognitive Status (TICS). Used to measure cognitive status. For TICS - the minimum = 0 maximum = 50. Higher scores mean better cognition.
Time Frame: Baseline prior to the workshop, at 3 months after baseline and at 6 months after baseline
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WW Treatment Group | WW Control Group
Number analyzed (Participants) | 130 | 123
score on a scale
  3 Months | .96 (4.02) | .92 (4.17)
  6 Months: number analyzed (Participants) | 123 | 122
  6 Months | 1.42 (4.15) | 1.22 (4.21)

3. Secondary Outcome: Change in Social Satisfaction
Description: Social Provisions Scale. Range of total score should be 24-96 with higher scores being a better outcome.
Time Frame: Baseline prior to the workshop, at 3 months after baseline and at 6 months after baseline
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WW Treatment Group | WW Control Group
Number analyzed (Participants) | 130 | 123
score on a scale
  3 Months | .30 (5.72) | -.72 (5.86)
  6 Months: number analyzed (Participants) | 123 | 122
  6 Months | 0.23 (12.69) | -.43 (12.79)

4. Secondary Outcome: Change in Physical Activity Levels
Description: Physical Activity Scale for the Elderly (PASE). Scores range from 0 to 793, with higher scores indicating greater physical activity
Time Frame: Baseline prior to the workshop, at 3 months after baseline and at 6 months after baseline
Population: Number analyzed changes due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WW Treatment Group | WW Control Group
Number analyzed (Participants) | 152 | 133
score on a scale
  Baseline | 68.21 (50.3) | 71.29 (63.85)
  3 Months: number analyzed (Participants) | 130 | 123
  3 Months | 57.34 (43.05) | 64.84 (60.41)
  6 Months: number analyzed (Participants) | 123 | 122
  6 Months | 68.35 (48.37) | 66.95 (35.0)

5. Secondary Outcome: Stress
Description: Perceived Stress Scale (PSS). Total scores range from 0 to 40. Higher scores indicate higher stress.
Time Frame: Baseline prior to the workshop, at 3 months after baseline and at 6 months after baseline
Population: Sample sizes change by time point due to loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WW Treatment Group | WW Control Group
Number analyzed (Participants) | 152 | 133
score on a scale
  Baseline | 21 (3.89) | 20.62 (3.5)
  3 Months: number analyzed (Participants) | 130 | 123
  3 Months | 19.94 (3.31) | 20.26 (3.34)
  6 Months: number analyzed (Participants) | 123 | 122
  6 Months | 19.65 (3.26) | 20.34 (3.89)

6. Secondary Outcome: Change in Sleep
Description: Pittsburgh Sleep Quality Index (PSQI). The PSQI has 7 sections which are scored. The seven component scores are then summed to yield a global PSQI score, which has a range of 0-21; higher scores indicate worse sleep quality.
Time Frame: Baseline prior to the workshop, at 3 months after baseline and at 6 months after baseline
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | WW Treatment Group | WW Control Group
Number analyzed (Participants) | 130 | 123
score on a scale
  3 Months | 0.21 (1.82) | -.17 (1.77)
  6 Months: number analyzed (Participants) | 123 | 122
  6 Months | 7.23 (2.51) | -6.37 (2.38)

7. Secondary Outcome: Self-efficacy
Description: PROMIS general self efficacy short-form. Survey scores are changed into a T score, with a mean of 50 and a standard deviation of 10. The higher the score the greater the self-efficacy.
Time Frame: Baseline prior to the workshop, at 3 months after baseline and at 6 months after baseline
Population: Sample size varies by time point due to drop out/loss to follow up.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | WW Treatment Group | WW Control Group
Number analyzed (Participants) | 152 | 133
T-score
  Baseline | 46.89 (8.00) | 49.61 (8.93)
  3 Months: number analyzed (Participants) | 130 | 123
  3 Months | 48.10 (8.47) | 50.22 (8.33)
  6 Months: number analyzed (Participants) | 123 | 122
  6 Months | 50.49 (8.48) | 49.28 (7.97)

ADVERSE EVENTS:
Time Frame: Enrollment through 6 month follow-up time point.
Arm/Group | WW Treatment Group | WW Control Group
All-Cause Mortality (participants affected / at risk) | 1/152 | 0/133
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/133
Other Adverse Events (participants affected / at risk) | 0/152 | 0/133

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT04928885/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT04928885/ICF_001.pdf